CLINICAL TRIAL: NCT03812029
Title: A Phase 2a, Randomized, Double-Blind, Multicenter, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of EYP001a in Patients With Nonalcoholic Steatohepatitis
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of EYP001a in Patients With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EYP001-202; 2018-003119-22 (EudraCT Number)
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: EYP001 (vonafexor); Liver Diseases; Non-alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Vonafexor 100 mg BID (Experimental): Oral dose twice daily for 12 weeks (84 days)
  Interventions: Drug: Vonafexor
- Vonafexor 200 mg QD (Experimental): Oral dose once daily for 12 weeks (84 days)
  Interventions: Drug: Vonafexor
- Vonafexor 400 mg QD (Experimental): Oral dose once daily for 12 weeks (84 days)
  Interventions: Drug: Vonafexor
- Placebo (Placebo Comparator): Oral dose twice daily for 12 weeks (84 days)
  Interventions: Other: Placebo
- Vonafexor 100 mg QD (Experimental): Oral dose once daily for 12 weeks (84 days)
  Interventions: Drug: Vonafexor

INTERVENTIONS:
Drug: Vonafexor — Oral tablets
  Arms: Vonafexor 100 mg BID; Vonafexor 100 mg QD; Vonafexor 200 mg QD; Vonafexor 400 mg QD
Other: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of EYP001a (Vonafexor) with respect to safety, tolerability, pharmacokinetics and on markers of liver inflammation in patients with NASH

DETAILED DESCRIPTION:
This is a 2-part, randomized, double-blind, multicenter, placebo-controlled study to evaluate the safety and efficacy of Vonafexor in patients with NASH who likely have stage F2 to F3 fibrosis at approximately 50 global clinical sites. Overall, approximately 114 eligible patients will be enrolled: 24 patients in Part A (Safety Run-in Cohort), followed by 90 patients in Part B.

In Part A, 24 patients will be randomized on Day 1 to 1 of 4 parallel treatment groups: 100 mg Vonafexor twice daily (BID), 200 mg Vonafexor once daily (QD), 400 mg Vonafexor QD, or placebo BID. In Part B, 90 patients will be randomized on Day 1 to 1 of 3 parallel treatment groups: 100 mg Vonafexor QD, 200 mg Vonafexor QD, or placebo QD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Suspected diagnosis of NASH, evidenced by elevated alanine aminotransferase (ALT), liver stiffness compatible with F2 or F3 fibrosis and Liver Fat Content (LFC) ≥10% as measured by MRI
* Women of childbearing potential and male patients with female partners must agree to use a dual method of contraception

Exclusion Criteria:

* Evidence of worsening liver injury
* Previous diagnosis of other forms of non-NASH liver disease
* Use of Vitamin E, glitazones, glucagon-like Peptide-1 receptor agonists, ursodeoxycholic acid, or obeticholic acid within 90 days prior to screening
* History of cirrhosis or liver decompensation
* Known history of alcohol abuse or daily heavy alcohol consumption
* Pregnant or breastfeeding women
* Type 1 diabetes mellitus and uncontrolled type 2 diabetes mellitus
* Patients with contraindications to MRI imaging

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Stephen, MD, Principal Investigator — Pinnacle Clinical Research
Locations (42):
- United States (24):
  - ENYO PHARMA Investigative site 0424, North Little Rock, Arkansas
  - ENYO PHARMA Investigative site 0418, Lakewood Rch, Florida
  - ENYO PHARMA Investigative site 0402, Ocoee, Florida
  - ENYO PHARMA Investigative site 0420, Orlando, Florida
  - ENYO PHARMA Investigative site 0419, Port Orange, Florida
  - ENYO PHARMA Investigative site 0403, Athens, Georgia
  - ENYO PHARMA Investigative site 0423, Savannah, Georgia
  - ENYO PHARMA Investigative site 0407, Snellville, Georgia
  - ENYO PHARMA Investigative site 0409, Indianapolis, Indiana
  - ENYO PHARMA Investigative site 0413, Baton Rouge, Louisiana
  - ENYO PHARMA Investigative site 0404, Marrero, Louisiana
  - ENYO PHARMA Investigative site 0422, Baltimore, Maryland
  - ENYO PHARMA Investigative site 0412, Jackson, Mississippi
  - ENYO PHARMA Investigative site 0414, Kansas City, Missouri
  - ENYO PHARMA Investigative site 0406, Durham, North Carolina
  - ENYO PHARMA Investigative site 0411, Columbus, Ohio
  - ENYO PHARMA Investigative site 0401, Charleston, South Carolina
  - ENYO PHARMA Investigative site 0408, Charleston, South Carolina
  - ENYO PHARMA Investigative site 0421, Rapid City, South Dakota
  - ENYO PHARMA Investigative site 0405, Arlington, Texas
  - ENYO PHARMA Investigative site 0416, Austin, Texas
  - ENYO PHARMA Investigative site 0417, Edinburg, Texas
  - ENYO PHARMA Investigative site 0410, San Antonio, Texas
  - ENYO PHARMA Investigative site 0415, San Antonio, Texas
- Belgium (4):
  - ENYO PHARMA Investigative site 0105, Brussels
  - ENYO PHARMA Investigative site 0101, Edegem
  - ENYO PHARMA Investigative site 0104, Ghent
  - ENYO PHARMA Investigative site 0103, Ghent
- France (8):
  - ENYO PHARMA Investigative site 0201, Angers
  - ENYO PHARMA Investigative site, Créteil
  - ENYO PHARMA Investigative site 0203, Limoges
  - ENYO PHARMA Investigative site 0204, Lyon
  - ENYO PHARMA Investigative site 0206, Paris
  - ENYO PHARMA Investigative site 0202, Pessac
  - ENYO PHARMA Investigative site 0207, Toulouse
  - ENYO PHARMA Investigative site 0205, Villejuif
- ENYO PHARMA Investigative site 0429, San Juan, Puerto Rico
- United Kingdom (5):
  - ENYO PHARMA Investigative site 0304, Belfast
  - ENYO PHARMA Investigative site 0302, Cambridge
  - ENYO PHARMA Investigative site 0303, London
  - ENYO PHARMA Investigative site 0305, London
  - ENYO PHARMA Investigative site 0301, Nottingham

REFERENCES:
- [Derived] Ratziu V, Harrison SA, Loustaud-Ratti V, Bureau C, Lawitz E, Abdelmalek M, Alkhouri N, Francque S, Girma H, Darteil R, Couchoux H, Wolf M, Sanyal A, Vonderscher J, Scalfaro P. Hepatic and renal improvements with FXR agonist vonafexor in individuals with suspected fibrotic NASH. J Hepatol. 2023 Mar;78(3):479-492. doi: 10.1016/j.jhep.2022.10.023. Epub 2022 Nov 9. PMID 36334688

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For Part A, data from the 3 vonafexor treatment groups were pooled and summarized. Due to the small number of subjects by treatment group in Part A, and as the Study EYP001 202 Part A Pharmacokinetic (PK) results between groups were found to be nonlinear with similar exposure for the vonafexor 200 mg once daily (QD) and vonafexor 400 mg QD groups, only the pooled vonafexor treatment group were compared with the placebo group.
Groups:
- Placebo Part A: Oral dose twice daily for 12 weeks (84 days)
  Placebo: Oral tablets
- Vonafexor Pooled Part A: Oral dose once or twice a day according to treatment arm for 12 weeks (84 days)
  Vonafexor: Oral tablets
- Placebo Part B: Oral dose once daily for 12 weeks (84 days)
  Placebo: Oral tablets
- Vonafexor 100 mg QD Part B; Vonafexor 200 mg QD Part B: Oral dose once daily for 12 weeks (84 days)
  Vonafexor: Oral tablets
Period: Overall Study
Arm/Group | Placebo Part A | Vonafexor Pooled Part A | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B
Started | 7 | 17 | 32 | 31 | 33
Completed | 5 | 7 | 32 | 25 | 23
Not Completed | 2 | 10 | 0 | 6 | 10
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 2
Not completed — Stopping rules | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 9 | 0 | 3 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: For Part A, data from the 3 vonafexor treatment groups were pooled and summarized. Due to the small number of subjects by treatment group in Part A, and as the Study EYP001 202 Part A PK results between groups were found to be nonlinear with similar exposure for the vonafexor 200 mg QD and vonafexor 400 mg QD groups, only the pooled vonafexor treatment group were compared with the placebo group.
Groups:
- Vonafexor Pooled Part A: Oral dose once or twice a day according to treatment arms for 12 weeks (84 days)
  Vonafexor: Oral tablets
- Total: Total of all reporting groups
Arm/Group | Placebo Part A | Vonafexor Pooled Part A | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B | Total
Number analyzed (Participants) | 7 | 17 | 32 | 31 | 33 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part A + Part B were analysed fully separately as per SAP and Study Protocol v5.0 with study populations slightly different between the 2 study parts.
  years
    Age Part A: number analyzed (Participants) | 7 | 17 | 0 | 0 | 0 | 24
    Age Part A | 48.7 (18.4) | 56.1 (8.9) |  |  |  | 54.0 (12.4)
    Age Part B: number analyzed (Participants) | 0 | 0 | 32 | 31 | 33 | 96
    Age Part B |  |  | 57.3 (10.3) | 58.1 (13.7) | 54.0 (11.9) | 56.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 14 | 18 | 14 | 21 | 69
  Male | 5 | 3 | 14 | 17 | 12 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 6 | 8 | 10 | 31
  Not Hispanic or Latino | 5 | 12 | 26 | 23 | 23 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 2 | 1 | 7
  White | 7 | 16 | 29 | 26 | 31 | 109
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 0 | 3
Height [Mean (Standard Deviation); unit: cm] — Population: Part A + Part B were analysed fully separately as per SAP and Study Protocol v5.0 with study populations slightly different between the 2 study parts.
  cm
    Height Part A: number analyzed (Participants) | 7 | 17 | 0 | 0 | 0 | 24
    Height Part A | 169.0 (7.4) | 163.2 (9.9) |  |  |  | 164.9 (9.5)
    Height Part B: number analyzed (Participants) | 0 | 0 | 32 | 31 | 33 | 96
    Height Part B |  |  | 168.1 (9.8) | 167.1 (8.5) | 166.8 (10.1) | 167.3 (9.4)
Weight [Mean (Standard Deviation); unit: kg] — Population: Part A + Part B were analysed fully separately as per SAP and Study Protocol v5.0 with study populations slightly different between the 2 study parts.
  kg
    Weight Part A: number analyzed (Participants) | 7 | 17 | 0 | 0 | 0 | 24
    Weight Part A | 112.4 (32.6) | 103.4 (25.4) |  |  |  | 106.0 (27.3)
    Weight Part B: number analyzed (Participants) | 0 | 0 | 32 | 31 | 33 | 96
    Weight Part B |  |  | 97.5 (18.3) | 95.8 (14.0) | 98.8 (18.4) | 97.4 (16.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Part A + Part B were analysed fully separately as per SAP and Study Protocol v5.0 with study populations slightly different between the 2 study parts.
  kg/m^2
    BMI Part A: number analyzed (Participants) | 7 | 17 | 0 | 0 | 0 | 24
    BMI Part A | 39.3 (10.2) | 38.8 (9.0) |  |  |  | 38.9 (9.1)
    BMI Part B: number analyzed (Participants) | 0 | 0 | 32 | 31 | 33 | 96
    BMI Part B |  |  | 34.3 (4.3) | 34.3 (4.1) | 35.4 (5.1) | 34.7 (4.5)
Waist circumference [Mean (Standard Deviation); unit: cm] — Population: Part A + Part B were analysed fully separately as per SAP and Study Protocol v5.0 with study populations slightly different between the 2 study parts.
  cm
    Waist circumference Part A: number analyzed (Participants) | 7 | 17 | 0 | 0 | 0 | 24
    Waist circumference Part A | 128.9 (31.5) | 116.1 (16.0) |  |  |  | 119.8 (21.7)
    Waist circumference Part B: number analyzed (Participants) | 0 | 0 | 32 | 31 | 33 | 96
    Waist circumference Part B |  |  | 112.6 (13.0) | 111.4 (8.6) | 114.1 (11.8) | 112.7 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Absolute Change From Baseline in Percentage of Fat in the Liver as Assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF)
Description: The liver fat percentage was assessed by MRI-PDFF, which is an established method that enables the quantification of fat content in the liver; the value of liver fat is expressed in percentage and ranges from 0 to 100% with higher values representing higher liver fat level.
Time Frame: 12 weeks
Population: For Part A, as per ICH, analysis were performed as defined in the SAP: data from the 3 vonafexor treatment groups were pooled and compared with the placebo group.
  The modified ITT (mITT) Population which was defined as patients from the ITT Population who have valid baseline and Week 12/Early Termination (ET) MRI-PDFF measurements of Liver Fat Content (LFC) has been used to analyse this endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of liver fat change
Arm/Group | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B | Placebo Part A | Vonafexor Pooled Part A
Number analyzed (Participants) | 32 | 28 | 28 | 5 | 12
Percentage of liver fat change | -2.3 [-4.0 to -0.6] | -6.3 [-8.1 to -4.5] | -5.4 [-7.2 to -3.6] | 3.9 [-2.5 to 10.4] | -4.7 [-8.5 to 0.9]
Statistical Analysis 1: Comparison: Placebo Part B vs Vonafexor 100 mg QD Part B; Test type: Superiority; p = 0.0015, ANCOVA — a priori threshold for statistical significance : <0.05
Statistical Analysis 2: Comparison: Placebo Part B vs Vonafexor 200 mg QD Part B; Test type: Superiority; p = 0.0121, ANCOVA — a priori threshold for statistical significance : <0.05
Statistical Analysis 3: Comparison: Placebo Part A vs Vonafexor Pooled Part A; Test type: Superiority; p = 0.0371, ANCOVA — a priori threshold for statistical significance : <0.05

2. Secondary Outcome: Analysis of Change From Baseline in Glomerular Filtration rate_Part B
Time Frame: 12 weeks
Population: The Intent-to-Treat (ITT) Population, which was defined as all patients who were randomized and administered at least 1 dose of study drug was used to analyse this endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B
Number analyzed (Participants) | 32 | 31 | 33
mL/min/1.73m2 | -2.7 [-6.6 to 1.2] | 6.2 [1.9 to 10.2] | 3.2 [-1.2 to 7.7]
Statistical Analysis 1: Comparison: Placebo Part B vs Vonafexor 100 mg QD Part B; Test type: Superiority; p = 0.003, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 2: Comparison: Placebo Part B vs Vonafexor 200 mg QD Part B; Test type: Superiority; p = 0.04, Mixed Models Analysis — a priori threshold for statistical significance : <0.05

3. Secondary Outcome: Analysis of Percent Change (Relative) From Baseline in Percentage of Fat in the Liver as Assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF)
Description: as for outcome 1
Time Frame: 12 weeks
Population: For Part A, as per ICH, analysis were performed as defined in the SAP: data from the 3 vonafexor treatment groups were pooled and compared with the placebo group.
  The modified ITT (mITT) Population which was defined as patients from the ITT Population who have valid baseline and Week 12/ET MRI-PDFF measurements of LFC has been used to analyse this endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B | Placebo Part A | Vonafexor Pooled Part A
Number analyzed (Participants) | 32 | 28 | 28 | 5 | 12
Percent change | -10.5 [-19.0 to -2.0] | -30.4 [-39.4 to -21.3] | -25.3 [-34.3 to -16.2] | 11.7 [-28.5 to 51.9] | -25.0 [-48.4 to -1.5]
Statistical Analysis 1: Comparison: Placebo Part B vs Vonafexor 100 mg QD Part B; Test type: Superiority; p = 0.0017, ANCOVA — a priori threshold for statistical significance : <0.05
Statistical Analysis 2: Comparison: Placebo Part B vs Vonafexor 200 mg QD Part B; Test type: Superiority; p = 0.018, ANCOVA — a priori threshold for statistical significance : <0.05
Statistical Analysis 3: Comparison: Placebo Part A vs Vonafexor Pooled Part A; Test type: Superiority; p = 0.13, ANCOVA — a priori threshold for statistical significance : <0.05

4. Secondary Outcome: Analysis of Change From Baseline in Corrected T1 (CT1)
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Arm/Group | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B | Placebo Part A | Vonafexor Pooled Part A
Number analyzed (Participants) | 32 | 28 | 28 | 5 | 12
msec | -9.9 [-38.5 to 18.7] | -80.2 [-110.6 to -49.8] | -71.8 [-100.4 to -43.2] | 35.0 [-27.0 to 97.0] | -58.2 [-98.7 to -17.8]
Statistical Analysis 1: Comparison: Placebo Part B vs Vonafexor 100 mg QD Part B; Test type: Superiority; p = 0.001, ANCOVA — a priori threshold for statistical significance : <0.05
Statistical Analysis 2: Comparison: Placebo Part B vs Vonafexor 200 mg QD Part B; Test type: Superiority; p = 0.002, ANCOVA — a priori threshold for statistical significance : <0.05
Statistical Analysis 3: Comparison: Placebo Part A vs Vonafexor Pooled Part A; Test type: Superiority; p = 0.018, ANCOVA — a priori threshold for statistical significance : <0.05

5. Secondary Outcome: Analysis of Change From Baseline in Alanine Aminotransferase (ALT)
Time Frame: 12 weeks
Population: For Part A, as per ICH, analysis were performed as defined in the SAP: data from the 3 vonafexor treatment groups were pooled and compared with the placebo group.
  The ITT Population, defined as all patients who were randomized and administered at least 1 dose of study drug was used to analyse this endpoint but for this endpoint 1 patient in Vonafexor 200 mg QD part B arm was excluded because he experienced a serious transaminase increase due to previously undiagnosed auto-immune hepatitis.
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B | Placebo Part A | Vonafexor Pooled Part A
Number analyzed (Participants) | 32 | 31 | 32 | 7 | 17
U/L | -11.7 [-18.9 to -4.6] | -16.3 [-24.1 to -8.4] | -7.5 [-15.3 to 0.4] | -4.1 [-27.5 to 19.3] | 17.7 [1.9 to 33.5]
Statistical Analysis 1: Comparison: Placebo Part B vs Vonafexor 100 mg QD Part B; Test type: Superiority; p = 0.09, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 2: Comparison: Placebo Part B vs Vonafexor 200 mg QD Part B; Test type: Superiority; p = 0.47, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 3: Comparison: Placebo Part A vs Vonafexor Pooled Part A; Test type: Superiority; p = 0.14, Mixed Models Analysis — a priori threshold for statistical significance : <0.05

6. Secondary Outcome: Analysis of Change From Baseline in Gamma Glutamyltranspeptidase (GT)
Time Frame: 12 weeks
Population: For Part A, as per ICH, analysis were performed as defined in the SAP: data from the 3 vonafexor treatment groups were pooled and compared with the placebo group.
  The Intent-to-Treat (ITT) Population, which was defined as all patients who were randomized and administered at least 1 dose of study drug was used to analyse this endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B | Placebo Part A | Vonafexor Pooled Part A
Number analyzed (Participants) | 32 | 31 | 33 | 7 | 17
U/L | -3.9 [-9.9 to 2.2] | -40.6 [-47.1 to -34.0] | -34.1 [-40.6 to -27.7] | 3.7 [-7.8 to 15.2] | -25.2 [-34.2 to -16.3]
Statistical Analysis 1: Comparison: Placebo Part B vs Vonafexor 100 mg QD Part B; Test type: Superiority; p < 0.0001, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 2: Comparison: Placebo Part B vs Vonafexor 200 mg QD Part B; Test type: Superiority; p < 0.0001, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 3: Comparison: Placebo Part A vs Vonafexor Pooled Part A; Test type: Superiority; p = 0.0002, Mixed Models Analysis — a priori threshold for statistical significance : <0.05

7. Secondary Outcome: Analysis of Change From Baseline in Body Weight
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B | Placebo Part A | Vonafexor Pooled Part A
Number analyzed (Participants) | 32 | 31 | 33 | 7 | 17
kg | -0.1 [-1.0 to 0.9] | -1.7 [-2.7 to -0.7] | -2.5 [-3.5 to -1.5] | 1.2 [-1.0 to 3.4] | -2.2 [-3.7 to -0.7]
Statistical Analysis 1: Comparison: Placebo Part B vs Vonafexor 100 mg QD Part B; Test type: Superiority; p = 0.017, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 2: Comparison: Placebo Part B vs Vonafexor 200 mg QD Part B; Test type: Superiority; p = 0.0006, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 3: Comparison: Placebo Part A vs Vonafexor Pooled Part A; Test type: Superiority; p = 0.006, Mixed Models Analysis — a priori threshold for statistical significance : <0.05

8. Secondary Outcome: Analysis of Change From Baseline in Waist Circumference
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B | Placebo Part A | Vonafexor Pooled Part A
Number analyzed (Participants) | 32 | 31 | 33 | 7 | 17
cm | 0.1 [-1.2 to 1.3] | -1.2 [-2.6 to 0.1] | -2.2 [-3.6 to -0.9] | -1.8 [-5.0 to 1.4] | -2.9 [-5.0 to -0.7]
Statistical Analysis 1: Comparison: Placebo Part B vs Vonafexor 100 mg QD Part B; Test type: Superiority; p = 0.16, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 2: Comparison: Placebo Part B vs Vonafexor 200 mg QD Part B; Test type: Superiority; p = 0.01, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 3: Comparison: Placebo Part A vs Vonafexor Pooled Part A; Test type: Superiority; p = 0.57, Mixed Models Analysis — a priori threshold for statistical significance : <0.05

9. Secondary Outcome: Analysis of Change From Baseline in Waist to Hip ratio_Part B
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: ratio
Arm/Group | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B
Number analyzed (Participants) | 32 | 31 | 33
ratio | 0.014 [0.001 to 0.026] | -0.017 [-0.031 to -0.003] | -0.010 [-0.024 to 0.004]
Statistical Analysis 1: Comparison: Placebo Part B vs Vonafexor 100 mg QD Part B; Test type: Superiority; p = 0.0017, Mixed Models Analysis — a priori threshold for statistical significance : <0.05
Statistical Analysis 2: Comparison: Placebo Part B vs Vonafexor 200 mg QD Part B; Test type: Superiority; p = 0.0093, Mixed Models Analysis — a priori threshold for statistical significance : <0.05

10. Secondary Outcome: Analysis of Change From Baseline in Glomerular Filtration rate_Part A
Description: For Part A, as per ICH, analysis were performed as defined in the SAP: data from the 3 vonafexor treatment groups were pooled and compared with the placebo group.
Time Frame: 12 weeks
Measure: Geometric Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo Part A | Vonafexor Pooled Part A
Number analyzed (Participants) | 7 | 17
mL/min/1.73m^2 | -4 (18.4) | -11.3 (12.5)

ADVERSE EVENTS:
Time Frame: After dose the first dose of study drug until D96
Groups:
- Vonafexor 100 mg BID Part A: Oral dose twice daily for 12 weeks (84 days)
  Vonafexor: Oral tablets
- Vonafexor 200 mg QD Part A; Vonafexor 400 mg QD Part A; Vonafexor 100 mg QD Part B; Vonafexor 200 mg QD Part B: Oral dose once daily for 12 weeks (84 days)
  Vonafexor: Oral tablets
Arm/Group | Placebo Part A | Vonafexor 100 mg BID Part A | Vonafexor 200 mg QD Part A | Vonafexor 400 mg QD Part A | Placebo Part B | Vonafexor 100 mg QD Part B | Vonafexor 200 mg QD Part B
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/5 | 0/6 | 0/32 | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/5 | 0/6 | 1/32 | 1/31 | 2/33
Other Adverse Events (participants affected / at risk) | 4/7 | 6/6 | 4/5 | 6/6 | 22/32 | 25/31 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Part A (N=7) | Vonafexor 100 mg BID Part A (N=6) | Vonafexor 200 mg QD Part A (N=5) | Vonafexor 400 mg QD Part A (N=6) | Placebo Part B (N=32) | Vonafexor 100 mg QD Part B (N=31) | Vonafexor 200 mg QD Part B (N=33)
Angina instable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Part A (N=7) | Vonafexor 100 mg BID Part A (N=6) | Vonafexor 200 mg QD Part A (N=5) | Vonafexor 400 mg QD Part A (N=6) | Placebo Part B (N=32) | Vonafexor 100 mg QD Part B (N=31) | Vonafexor 200 mg QD Part B (N=33)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electric shock (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (4) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (7) | 4 (5) | 6 (10) | 4 (4) | 19 (29) | 22 (36)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data may be considered for publication in a scientific journal or for reporting at a scientific meeting. Each Investigator is obligated to keep data pertaining to the study confidential. The Investigator must consult with the Sponsor before any study data are submitted for publication. The Sponsor reserves the right to deny publication rights until mutual agreement on the content, format, interpretation of data in the manuscript, and journal selected for publication are achieved.

DOCUMENTS (2):
  • Study Protocol (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT03812029/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT03812029/SAP_001.pdf